CLINICAL TRIAL: NCT00990977
Title: A Prospective, Randomized Controlled Trial of Mindfulness-based Stress Reduction (MBSR) Among Women Operated for Breast Cancer
Brief Title: Mindfulness and Cancer Mamma - Clinical Trial MBSR Among Women Operated for Breast Cancer
Acronym: MICA
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Danish Cancer Society (Other)
Collaborators: University of Copenhagen (Other); Herlev Hospital (Other)
Responsible Party: Principal Investigator, Trille Kjær, Ph.d-fellow, Danish Cancer Society
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DanishCS; 2007-41-1654 (Registry Identifier: Danish Data Protection Agency)
Record Dates: First submitted 2009-10-02; First posted 2009-10-07 (Estimated); Last update posted 2015-06-30 (Estimated); Status verified 2015-06

CONDITIONS: Breast Cancer
Keywords: breast cancer; supportive care; post-treatment; intervention; MBSR; mindfulness; anxiety; depression; lifestyle; diet; alcohol consumption; smoking; exercise; spirituality; existential well-being; physical symptoms; women
MeSH Terms: conditions — Breast Neoplasms; Anxiety Disorders; Depression; Alcohol Drinking; Smoking; Motor Activity | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- controls (No Intervention): assessment only
- cases (Experimental): MBSR including brief information session and assessments
  Interventions: Behavioral: mindfulness based stress reduction (MBSR)

INTERVENTIONS:
Behavioral: mindfulness based stress reduction (MBSR) — MBSR is an 8-week course covering a total of 24 contact hours where the group of patients meet with an clinical psychologist certified as mindfulness instructor. The group will train the ability of mindfulness by specific awareness improving practises (body-scan) guided meditations and soft yoga. Between group-sessions participants are recommended to practice 45 minutes daily and to go through instructions in MBSR hand-outs. Participants will be given audio-CDs containing instructions and guides to support home practice.
  Other Names: MBSR (Kabat-Zinn)
  Arms: cases

SUMMARY:
The number of Danish women treated for breast cancer rise every year, though survival rates have improved, women can still expect to experience the diverse late effects reported by this group of patients. Mindfulness labels the ability to be aware of the present moment - thereby avoiding speculations about both past and present. Mindfulness based stress-reduction (MBSR) is an 8-week program, covering 24 contact-hours and 45 minutes daily home practice. The program aims at developing participants' coping resources and developing participants' mindful awareness. Thus the program consists of guided meditations, guided body scan(a specific awareness exercise)and through meditation, yoga and psychoeducation concerning stress and stress-reactions, while meditation and bodyscan is practiced at home by the use of specific audio-CDs guiding the patient. The MBSR-program have shoved promising results among patients with anxiety-disorders, depression and chronic pain. Smaller studies have also found positive effects of the program among cancer patients. The investigators want to evaluate the effect of the MBSR program on levels of anxiety and depression as well as the possible influence of mindfulness training on health behaviors and existential concerns. The study are based on the following hypotheses:

* report of anxiety and depression will decrease among cases
* better compliance will lead to more decrease in levels of anxiety and depression
* cases will make lifestyle changes suitable with recommendations for BC patients in post-treatment phase of the illness
* decreased level of anxiety and depression will reflect improved spiritual well-being
* improved spiritual wellbeing will lead to decreased report of physical symptoms

All participants in this randomized controlled trial will fill out questionnaires at enrollment and as 1, 6 and 12 months follow-up. Based on results from this trial clinicians and patients will be able to make decisions regarding post-treatment psychosocial intervention and researchers will have initial evidence of the effect of the intervention and thus possible indications for research on mindfulness among patients diagnosed with cancer at other stages or sites.

DETAILED DESCRIPTION:
Original Research Protocol, Copenhagen January 2007 Cancer and Mindfulness: A prospective, randomized trial of a psychosocial intervention among women operated for breast cancer

Background From the time of diagnosis cancer patients have a need for psychological support. Many patients handle the situation by the help of friends and family, while others need professional support to come to terms with different phases of life as a cancer patient. Only few randomized trials have been conducted in order to determine what kinds of professional support patients will benefit from. These studies conclude that the prevalence of anxiety and depression in reduced. This is of major importance as depending of cancer type, treatment modality, age and gender, a total of 10-50 % of Danish cancer patients reports such well-defined psychosocial symptoms following the diagnosis of cancer.

Mindfulness meditation aims to increase the experience of presence and an increased relation to several emotional and sensory experiences. Instead of being a technique aimed to control and change unwanted psychological states the method is rather a way to stay present in the here and now without judging and as such it has been developed into a stress reduction method: mindfulness based stress reduction (MBSR). The method is taught within a group setting by an instructor guiding the patients during a week long program. The method has been evaluated within a variety of settings and has been found to effectively reduce symptoms related to different stress and pain conditions i.e. psoriasis, chronic pain, HIV/AIDS, anxiety and depression.2 Based on these experiences several programs have been developed and the program developed by Williams and Kabatt-Zinn has gained status as the most commonly applied and best validated. Within recent years the program has been included into cognitive-behavioral therapy. But with potential effects not only as reduction of symptoms but further opens the opportunity for participants to approach spiritual and existential themes. The potential effect is therefore not limited to simple reduction of symptoms but includes increased meaningfulness, quality of life and sense of coherence.

Nine studies of the effect of MBSR haw been conducted, including 10- 157 adult cancer patients being taught MBSR in groups of mainly breast cancer patients, but only three of these trials have been conducted as randomized controlled trials. I these trials patients have self-referred (selection bias), analysis have not been adjusted for biological status of the cancer disease (confounding), samples have been small (n=10-157) (type 2 error) and patients have differed with regard to time since diagnosis (misclassification). Despite these methodological limitations a tendency of positive effects of MBSR participation on psychological and physiological outcomes has been observed.

Yet it is still not determined whether MBSR will provide cancer patients benefit improving their daily life with cancer. Some important aspects have not been addressed in previous studies: When MBSR is applied as an intervention dose-response relation has only been observed among patients with a moderate level of symptoms. Thus sensitivity of MBSR in relation to stages of cancer, levels of pain or negative effects of treatments. We still do not know whether all cancer patients will profit from this type of intervention. Further the influence of patient compliance and working alliance is still not explored.

The diagnosis of cancer accentuates existential dimensions as spirituality and quality of life. Yet we do not know how MBSR can support patients in dealing with such themes. Be review of literature regarding patients coping with cancer the patients demand for interventions supporting their need to deal with existential themes is striking.

Aim We will conduct a randomized controlled trial among women diagnosed with primary breast cancer in order to evaluate the effect of MBSR on depression, anxiety quality of life, health behavior and psychological well-being.

Research questions

* We do not know whether all types of cancer patients will benefit from MBSR. Especially patients compliance must be empirically documented
* Cancer accentuates an array of existential concerns and the effect of MBSR on these subjective concerns must be examined

Inclusion All patient diagnosed with primary breast cancer in Department of Breast Surgery, Copenhagen Hospital Herlev, will be invited to participate in the study and in the randomization allocating patients to either MBSR intervention or treatment as usual control. Patients diagnosed and in active treatment for major psychiatric disease, patients with musculoskeletal disease and cardiovascular disease hindering MBSR participation, and patients previously diagnosed with other cancers than non-melanoma skin cancer will be excluded. A project nurse will contact eligible patients, deliver oral and written information and collect informed consent. If the patient consents baseline questionnaire will be administered.

Randomization will then take place. The project nurse will up-load patient data on secured project home-page. Computer generated sequence will automatically assign a unique study number to each patient indicating which study group she is allocated to. Result of the randomization will be delivered to the patient by the project nurse and potential disappointment will be handles at this point, and information regarding optional counseling provided by the Danish Cancer Society will also be given.

Intervention group MBSR will be delivered in groups of maximum 20 participants. The course will follow an 8 week schedule with 2-2½ hour sessions each week and instruction to practice 45 minutes daily at home. Upon conclusion of the course each group will participate in a full-day course (8 hours). The courses will be delivered by a manual (including audio CDs) developed by Antonia Sumbundu (see attached file). The group must meet in a quiet room large enough to room 20 persons lying down, as well as mats, carpets and chairs. The courses will be delivered in locations not affiliated with a hospital.

Control group The control group will receive treatment as usual and thus follow the standard control program applied by the surgical department.

* Questionnaire Prior to randomization and as follow-up after 6 and 12 months both study groups will be mailed questionnaires containing validated psychometric
* Hospital charts Descriptions of breast cancer operation, pathology of tumor as well as day to day entries will be collected.
* Administrative registries Data regarding comorbidity of all eligible patients will be collected in National Patient Registry and Central Psychiatric Registry upon finalization of the project.
* Qualitative outcomes Data collected by standardized self-report instruments will be supplemented by qualitative interviews inviting the intervention group participants to present themselves by giving an account of the treatment and a personal evaluation of the potential benefit.

Analysis

* Quantitative data Data will be stores in a database at the institute. Logistic regression analysis will be applied to evaluate which background variables effects participation. Analysis of outcomes will be conducted by applying multiple regressions at each time point. For simultaneous analysis of all follow-up times a linear mixed model with random effects of persons will be fitted. Outcomes as relapse and death among intervention group in comparison to both control group and non-participants will be analyzed by use of Cox regression model, controlling for the effect of biological and demographic variables. Analysis will be conducted under supervision of a senior statistician at the Department of Statistics and Epidemiology at the Institute.
* Qualitative data Based on the qualitative interviews a set of data-driven categories will be developed. These categories will be quantitatively evaluated. The transcript of the patient's self-presentation (approximately 2 pages) will be analyzed by use of qualitative methods, allowing for grouping of content categories as expressed by the patients. Statistical analysis will be applied to evaluate these categories.

Ethics Application of permission to conduct the study will be submitted to the The National Committee on Health Research Ethics and to the Danish Data Protection Agency. In information to patients regarding the study it will be stressed that participation is voluntary and that patients withdraw without any explanation at any time, and that withdrawal will have no influence on treatments delivered. Both written and oral consent must be given prior to participation. A short report will be mailed to all participants upon conclusion of the study. Vital status of participants will be checked in Central Persons Registry prior to any sending of study questionnaire. Data kept in the study database will be encrypted ensuring that only authorized scientific staff will be able to identify individuals. The encryption code will be kept by study manager. Results will be reported as tables and figures hindering identification of individuals. Also in the reporting of qualitative data will the quoted participants be kept anonymous.

Reference List

1. Ross L, Boesen E, Dalton S, Johansen C. Mind and cancer: does psychological intervention improve suvival and psychological well-being? European Journal of Cancer 2001.
2. Ott MJ, Norris RL, Bauer-Wu SM. Mindfulness meditation for oncology patients: a discussion and critical review. Integr Cancer Ther 2006; 5(2):98-108.
3. Bower JE, Ganz PA, Desmond KA, Rowland JH, Meyerowitz BE, Belin TR. Fatigue in Breast Cancer Survivors: Occurrence, Correlates, and Impact on Quality of Life. J Clin Oncol 2000; 18(4):743.
4. Bower JE, Ganz PA, Desmond KA et al. Fatigue in long-term breast carcinoma survivors: a longitudinal investigation. Cancer 2006; 106(4):751-758.

ELIGIBILITY:
Inclusion Criteria:

* women 18-75 years
* operated for breast cancer stage I-III at either Herlev hospital (F-118) or Ringsted sygehus (Mammakirurgisk Klinik) after september 2006
* speak and read danish

Exclusion Criteria:

* other cancers
* diseases or disabilities hindering MBSR-participation
* active treatment for psychiatric disease including alcohol abuse

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Actual)
Dates: Start 2008-03; Primary Completion 2010-12 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
SCL-90r Depression and anxiety subscales | baseline - 12 months

SECONDARY OUTCOMES:
clinical databases, containing information on BC (stage, treatment protocol) and comorbidity (other acute or chronic physical or psychiatric diseases) | baseline - 12 months
standardized validated psychometric scales | baseline - 12 months
  SCL-90r, NEO-PIR, FACIT-Sp, CES-D,MDI, WHO5, Inter99, IPAQ, FFMQ, BCPT-BEES,

CONTACTS AND LOCATIONS:
Overall Officials: Christoffer Johansen, M.D., Ph.D., Study Chair — Head Survivorship, Danish Cancer Society Research Center
Locations (1):
- Danish Cancer Sociaty Research Center, Suvivorship, Copenhagen, Ø, Denmark

REFERENCES:
- [Derived] Wurtzen H, Dalton SO, Christensen J, Andersen KK, Elsass P, Flyger HL, Pedersen AE, Sumbundu A, Steding-Jensen M, Johansen C. Effect of mindfulness-based stress reduction on somatic symptoms, distress, mindfulness and spiritual wellbeing in women with breast cancer: Results of a randomized controlled trial. Acta Oncol. 2015 May;54(5):712-9. doi: 10.3109/0284186X.2014.997371. Epub 2015 Mar 9. PMID 25752972
- [Derived] Jensen CG, Elsass P, Neustrup L, Bihal T, Flyger H, Kay SM, Khan S, Jensen SS, Pedersen A, Wurtzen H. What to listen for in the consultation. Breast cancer patients' own focus on talking about acceptance-based psychological coping predicts decreased psychological distress and depression. Patient Educ Couns. 2014 Nov;97(2):165-72. doi: 10.1016/j.pec.2014.07.020. Epub 2014 Jul 22. PMID 25086446
- [Derived] Andersen SR, Wurtzen H, Steding-Jessen M, Christensen J, Andersen KK, Flyger H, Mitchelmore C, Johansen C, Dalton SO. Effect of mindfulness-based stress reduction on sleep quality: results of a randomized trial among Danish breast cancer patients. Acta Oncol. 2013 Feb;52(2):336-44. doi: 10.3109/0284186X.2012.745948. Epub 2013 Jan 3. PMID 23282113
- [Derived] Wurtzen H, Dalton SO, Elsass P, Sumbundu AD, Steding-Jensen M, Karlsen RV, Andersen KK, Flyger HL, Pedersen AE, Johansen C. Mindfulness significantly reduces self-reported levels of anxiety and depression: results of a randomised controlled trial among 336 Danish women treated for stage I-III breast cancer. Eur J Cancer. 2013 Apr;49(6):1365-73. doi: 10.1016/j.ejca.2012.10.030. Epub 2012 Dec 19. PMID 23265707
- [Derived] Wurtzen H, Dalton SO, Andersen KK, Elsass P, Flyger HL, Sumbundu A, Johansen C. Who participates in a randomized trial of mindfulness-based stress reduction (MBSR) after breast cancer? A study of factors associated with enrollment among Danish breast cancer patients. Psychooncology. 2013 May;22(5):1180-5. doi: 10.1002/pon.3094. Epub 2012 May 16. PMID 22592966